CLINICAL TRIAL: NCT01487941
Title: Efficacy and Safety of the Setrox JS Lead (J=J-shaped, S=Screw)
Brief Title: Setrox JS Master Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 56
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is the evaluation of safety and efficacy of the pacemaker lead "Setrox JS".

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for pacemaker therapy
* Available for follow-up visits on a regular basis at the investigational site
* Contractual capability and ability to consent
* Age ≥18 years

Exclusion Criteria:

* Meet one or more of the contraindications for pacemaker therapy
* Permanent atrial fibrillation
* Have a life expectancy of less than six months
* Cardiac surgery in the next six months
* Enrolled in another cardiac clinical investigation
* Have other medical devices that may interact with the implanted pacemaker
* Pregnant and breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pacemaker indication
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Effect rate | 6 months
Atrial pacing threshold from Setrox JS at 3 month follow-up < 1.0V | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- SV. Anny Clinic Brno, Brno, Czechia